CLINICAL TRIAL: NCT01334125
Title: Glycemic Control in Children and Adolescents With Double Diabetes: Trial of Optimized Insulin-Metformin Regimen
Brief Title: Adjunctive Metformin Therapy in Double Diabetes
Acronym: AMTIDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Benjamin U. Nwosu, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13938
Record Dates: First submitted 2011-03-21; First posted 2011-04-12 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus
Keywords: Double Diabetes; Type 1 diabetes; Type 2 diabetes; Obesity; Acanthosis nigricans; Diabetes associated autoantibodies
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Obesity; Acanthosis Nigricans | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin 1000 mg once daily by mouth for 9 months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): 2 capsules once daily by mouth for 9 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 1000 mg once daily by mouth for 9 months
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — 2 capsules once daily by mouth for 9 months
  Arms: Placebo

SUMMARY:
The significance of this project is to investigate the effects of adjunctive metformin therapy in children and adolescents with double diabetes. Double diabetes describes a clinical state where an individual possesses features of both type 1 and type 2 diabetes. There is a paucity of data on the role of adjunctive metformin therapy in children and adolescents with double diabetes. To help fill this knowledge gap, the investigators propose a randomized, double-blind, placebo-controlled trial of metformin in double diabetes. Specifically, the investigators will evaluate changes in hemoglobin A1c and anthropometry in patients with a diagnosis of type 1 diabetes who also have features of type 2 diabetes or metabolic syndrome as well as patients with type 2 diabetes who possess diabetes-associated autoantibodies. This will help determine the safety profile, and efficacy of adjunctive metformin therapy in these subjects.

DETAILED DESCRIPTION:
In this 12-month clinical trial, a 3-month run-in period will precede the interventional phase of the study. All patients will be placed on treat-to-target insulin regimen alone during the run-in phase. At the end of the 3-month run-in period, all participants will continue on treat-to-target insulin regimen, and will then be randomized to either of the 2 arms of the study: an experimental arm, consisting of treat-to-target insulin regimen plus metformin, and a control arm consisting of treat-to-target insulin regimen plus placebo. Both the physicians and patients will be blinded to the oral agents being administered to patients.

ELIGIBILITY:
Inclusion Criteria:

A. General inclusion criteria

1. Ten to 20 years of age.
2. Pubertal (Tanner stages 2-5, by examination).
3. Hemoglobin A1c level of > 8.0% in the 6 months prior to enrollment.
4. All subjects must have access to a computer.

B. Specific inclusion criteria: [Subjects could have either #1, or #2].

1. Subjects with clinical and biochemical features of T2DM of > 6mo duration who also have positive T1DM antibodies

   * Clinical features: acanthosis nigricans, BMI >85%
   * Biochemical: evidence of insulin resistance at diagnosis
   * fasting insulin >27 uIU/mL(normal range 6-27) at a fasting blood glucose of ≥ 126 mg/dL, or
   * fasting c-peptide level of > 7.1 ng/mL (normal range 0.9 - 7.1), or
   * Homeostasis model of insulin resistance of >3.16
2. Patients with T1DM of > one yr duration with BMI >85%

   * Presentation with ketoacidosis at diagnosis
   * C-peptide <0.9 ng/mL (normal range 0.9 - 7.1),or (insulin < 6 uIU/mL) (NR 6-27) at diagnosis (when blood glucose is ≥ 126 mg/dL)
   * Can be antibody positive or negative
   * Increased insulin requirement (>2 Units/kg/day)

Exclusion Criteria:

1. Subjects on weight altering medications, such as orlistat.
2. Subjects with eating disorder
3. Subjects on medications other than insulin and or metformin that may affect blood glucose level.
4. Subjects with abnormal hepatic function tests.
5. Subjects with nephropathy, defined in this case as an overnight albumin excretion rate of >200 mcg/min using a first morning urine sample collection.
6. Subjects with recurrent diabetes ketoacidosis (more than 2 episodes in the past 12 months), or recurrent severe hypoglycemia (more than 2 episodes of hypoglycemia with altered level of consciousness, requiring assistance to treat in the past year).
7. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures.
8. Known or suspected allergy to metformin.
9. The receipt of any investigational drug within 6 months prior to this trial.
10. Active malignant neoplasms.
11. No access to a computer.
12. Subjects currently taking metformin for clinical purposes are not eligible to be enrolled in this study.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin U Nwosu, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UmassMemorial Medical Center, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Nwosu BU, Maranda L, Cullen K, Greenman L, Fleshman J, McShea N, Barton BA, Lee MM. A Randomized, Double-Blind, Placebo-Controlled Trial of Adjunctive Metformin Therapy in Overweight/Obese Youth with Type 1 Diabetes. PLoS One. 2015 Sep 14;10(9):e0137525. doi: 10.1371/journal.pone.0137525. eCollection 2015. PMID 26367281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a tertiary institution. The first patient was recruited on March 3rd 2011, and the last study patient was recruited on August 1, 2013. The study was closed on August 8, 2013.
Pre-assignment Details: Following enrollment, all subjects entered a run-in phase of 3-month duration during which participants were placed on insulin aspart and insulin detemir, and the treat-to-target insulin regimen (TTIR) started.
Groups:
- Placebo: 1 capsule once daily by mouth for 9 months
  Placebo: 1 capsule once daily by mouth for 9 months
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 15 | 13
Completed | 12 (3 subjects move to another city) | 10 (3 subjects left for college and moved out of the area)
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: Subjects who completed the baseline evaluation at the time of randomization were included in the baseline analysis.
Groups:
- Placebo: 1 capsule once daily by mouth for 9 months
  Placebo: 1 capsules once daily by mouth for 9 months
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (2.5) | 14.5 (3.1) | 14.7 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Baseline Adjusted Hemoglobin A1c Over Time
Description: Comparison of the baseline-adjusted differences in HbA1c between the metformin and placebo groups during the trial. Hemoglobin A1c is a marker of glycemic control. The reported values represented means adjusted for baseline values, age, gender, and BMI using repeated measures ANOVA (General Linear Model).
Time Frame: Baseline, 3mo, 6mo, and 9 months
Measure: Mean (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 15 | 13
percentage of HbA1c | 9.46 [8.47 to 10.46] | 9.85 [8.82 to 10.88]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Analyses were based on the intent-to-treat principle and were performed using SPSS v.22 (IBM Corporation, Armonk, NY); Test type: Superiority or Other; p = 0.903, ANOVA — Individual two-way mixed ANOVA models were fitted for each of our outcomes of interest, with treatment type (metformin or placebo) as the fixed effect, and baseline values, age, gender, and BMI as covariates

2. Secondary Outcome: Baseline Adjusted Changes in Lipid Profile Over Time
Description: Comparison of the baseline-adjusted differences in total cholesterol/high density cholesterol index over time between the metformin and the placebo groups. The reported values represented means adjusted for baseline values, age, gender, and BMI using repeated measures ANOVA (General Linear Model).
Time Frame: Baseline, 3mo, 6mo, and 9 months
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 15 | 13
ratio | 3.5 [3.0 to 4.1] | 4 [3.3 to 4.4]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Analyses were based on the intent-to-treat principle and were performed using SPSS v.22 (IBM Corporation, Armonk, NY); Test type: Superiority or Other; p = 0.578, ANOVA — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Baseline Adjusted Changes in Adiponectin/Leptin Ratio Over Time
Description: Comparison of the baseline-adjusted differences in adiponectin/leptin ratio over time between the metformin and the placebo groups. The reported values represented mean adjusted for baseline values, age, gender, and BMI using repeated measures ANOVA (General Linear Model).
Time Frame: Baseline, 3mo, 6 mo, and 9 months
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 15 | 13
ratio | 2.0 [0.84 to 3.2] | 1.2 [0.11 to 2.3]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Two way ANOVA comparison of the means of the adiponectin/leptin ratios between the metformin and placebo groups; Test type: Superiority or Other; p = 0.057, ANOVA

4. Secondary Outcome: Number of Participants With Minor, Major, and Nocturnal Hypoglycemia
Description: Comparison of the occurrence of hypoglycemic event requiring a third party assistance (major hypoglycemia) per subject during the study, and minor hypoglycemia (plasma glucose of <60 mg/dL or no measurement), as well as nocturnal hypoglycemia (plasma glucose of ≤60 mg/dL between 11PM and 6AM).
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 15 | 13
participants
  Major hypoglycemia | 1 | 0
  Minor hypoglycemia | 3 | 2
  Nocturnal hypoglycemia | 2 | 2
Statistical Analysis 1: Comparison: Metformin vs Placebo; p value represents the analysis for minor hypoglycemia; Test type: Superiority or Other; p = 1.00, t-test, 2 sided
Statistical Analysis 2: Comparison: Metformin vs Placebo; p value represents the analysis of the nocturnal hypoglycemia; Test type: Superiority or Other; p = 1.00, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 4/15 | 1/13
Other Adverse Events (participants affected / at risk) | 1/15 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=15) | Placebo (N=13)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Endocrine disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Severe hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=15) | Placebo (N=13)
Eye infection (Eye disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hidradenitis (Immune system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was stopped before reaching enrollment target because most youth were reluctant to commit to this long-term study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No